CLINICAL TRIAL: NCT04660448
Title: Lung Ultrasound Score and Pediatric Intensive Care Outcomes: a Prospective Observational Multicenter Study
Brief Title: Lung Ultrasound Score and Pediatric Intensive Care Outcomes (LUS-PICO)
Acronym: LUS-PICO
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Responsible Party: Sponsor
Other Study IDs: FINBA_CritLab_3
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Lung Injury; Extravascular Lung Water; Pulmonary Edema; Acute Respiratory Distress Syndrome; Shock
MeSH Terms: conditions — Lung Injury; Pulmonary Edema; Respiratory Distress Syndrome; Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bedside lung ultrasound examination — Lung ultrasound exploring 12 areas (6 in each lung) at 12 +/- 6 hours and at 48-72 hours from PICU admission. Clinical and analytical data collection coinciding with ultrasound imaging and during follow-up while admitted to PICU.

SUMMARY:
Bedside lung ultrasonography helps to obtain reliable clinical information about lung aeration, that has been categorized by means of the so-called lung ultrasound score (LUS). In critically ill adults, LUS has been related with the outcome both in patients with respiratory and some non-respiratory conditions. Pediatric studies about lung aeration have been done mainly on postoperative cardiac patients and infants with bronchiolitis. In this prospective, observational, multicenter, feasibility and diagnostic accuracy study, we will explore the degree of lung aeration impairment as a potential outcome predictor in critically ill children with a variety of underlying conditions. Children from 1 month to 18 years of age admitted to PICU will be recruited and LUS will be calculated at two time points: at 12 ± 6 hours and at 48-72 hours. Univariate and multivariate statistical analysis will be performed in order to ascertain the outcome influence of clinical factors in general and LUS in particular.

DETAILED DESCRIPTION:
Lung aeration can be assessed at the bedside by means of lung ultrasound, a non-invasive, quick, simple, and reproducible technique. It provides semiquantitative information about the amount of extravascular lung water (EVLW), which correlates with lung aeration. Accumulation of EVLW occurs secondarily to acute lung injury due to infection, inflammation or fluid overload. Lung aeration, measured by the lung ultrasound score (LUS), has been associated to patients' outcome in several studies in adult patients, suggesting that critically ill subjects showing higher degree of aeration loss have a worse outcome. This fact has been shown not only in patients with baseline respiratory conditions (for example in severe acute respiratory syndrome coronavirus 2), but also in adults with non-respiratory conditions, such as shock and in high-risk postoperative patients. Furthermore, animal studies have suggested that information obtained through lung ultrasonography may precede clinical signs and could help anticipate focused treatment.

To date, pediatric studies addressing the potential relationship between LUS and the outcome of critically ill children are scarce and limited to postoperative cardiac patients and infants with bronchiolitis.

In our research, children from 1 month to 18 years of age admitted to pediatric intensive care unit (PICU) who fulfill inclusion criteria will be recruited and will undergo point of care lung ultrasound examination at 12 ± 6 hours and at 48-72 hours from admission. Clinical data will be recorded and LUS will be calculated. The main objective of our study is to assess the potential role of LUS (as a semiquantitative indicator or lung aeration) as a feasible and reliable outcome prediction tool in children admitted to PICU. Secondary objectives will include to analyze the correlations between LUS and the need and length of ventilatory support, inflammatory and cardiac markers, hydric balance, renal replacement therapies requirement, and validated prognostic scales, as well as age, underlying disease, co-morbidities, length-of-stay, and other clinical characteristics of included children.

Patients with acute respiratory distress syndrome (ARDS) or shock during PICU admission time will also undergo additional lung ultrasound examinations at 12 ± 6 hours and at 48-72 hours from ARDS or shock diagnosis, as these subgroups represent a very specific and severe cohort of patients, which merits further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 month to 18 years-old admitted to PICU due to an acute condition

Exclusion Criteria:

1. - Children admitted to PICU to perform a procedure or to adjust a certain treatment (eg, home ventilatory support).
2. - Children with chronic pulmonary pathology (cystic fibrosis, bronchopulmonary dysplasia, etc…)
3. - Preoperative admissions in a stable condition (eg. Patient admitted previously to cardiac surgery)
4. - Inability to obtain interpretable ultrasonographic images due to bad ultrasonographic window
5. - Non disponibility of investigator
6. - High frequency ventilation
7. - Lack of clinical data

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 1 month to 18 years-old admitted to PICU due to an acute condition
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Requirement of invasive mechanical ventilation for more than 96 hours | 96 hours
  To evaluate the correlation of LUS obtained in the first 72 hours of admission with the need of invasive ventilatory support for over 96 hours. A comparison between patients with a respiratory condition versus non-respiratory condition as the cause of admission will be performed.

SECONDARY OUTCOMES:
Correlation between lung aeration and bedside inflammatory markers | 72 hours
  To evaluate the relation between lung aeration estimated by LUS and bedside inflammatory markers (C reactive protein, interleukin-6, procalcitonin, ferritin)
Correlation between lung aeration and bedside cardiac markers | 72 hours
  To evaluate the relation between lung aeration estimated by LUS and bedside cardiac markers (Brain natriuretic peptide, N-terminal proBNP, troponin, cystatin C)
Correlation between lung aeration and hydric balance and the need of renal replacement therapy | 72 hours
  To evaluate the relation between lung aeration estimated by LUS and hydric balance and the need of renal replacement therapy
Correlation between LUS and pediatric mortality scales | 72 hours
  To evaluate the relation between lung aeration and three prognostic indexes: pediatric risk of mortality (PRISM) III, pediatric sequential organ failure assessment (pSOFA), pediatric logistic organ dysfunction 2 (PELOD-2). It will also be assessed whether LUS may add any prognostic capacity to these scales.
Comparison of LUS calculation exploring 12 areas versus 8 areas | 72 hours
  To compare the prognostic ability of LUS calculated employing 12 lung zones versus LUS obtained using 8 zones (anterior and lateral areas exclusively)

OTHER OUTCOMES:
Utility of LUS in patients diagnosed with acute respiratory distress syndrome (ARDS) after 24 hours of admission | 72 hours
  All previously specified objectives will be evaluated in children diagnosed with ARDS. In those cases, LUS will be calculated at 12 +/- 6 hours and 72 hours from ARDS diagnosis.
Utility of LUS in patients diagnosed with shock after 24 hours of admission | 72 hours
  All previously specified objectives will be evaluated in children diagnosed with shock after 24 hours from admission. In those cases, LUS will be calculated at 12 +/- 6 hours and 72 hours from shock diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M. Albaiceta, MD PhD, Study Chair — HUCA-FINBA. Universidad de Oviedo; Juan Mayordomo-Colunga, MD PhD, Principal Investigator — HUCA-FIBA
Locations (1):
- Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh Y, Tissot C, Fraga MV, Yousef N, Cortes RG, Lopez J, Sanchez-de-Toledo J, Brierley J, Colunga JM, Raffaj D, Da Cruz E, Durand P, Kenderessy P, Lang HJ, Nishisaki A, Kneyber MC, Tissieres P, Conlon TW, De Luca D. International evidence-based guidelines on Point of Care Ultrasound (POCUS) for critically ill neonates and children issued by the POCUS Working Group of the European Society of Paediatric and Neonatal Intensive Care (ESPNIC). Crit Care. 2020 Feb 24;24(1):65. doi: 10.1186/s13054-020-2787-9. PMID 32093763
- [Background] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127
- [Background] Xirouchaki N, Kondili E, Prinianakis G, Malliotakis P, Georgopoulos D. Impact of lung ultrasound on clinical decision making in critically ill patients. Intensive Care Med. 2014 Jan;40(1):57-65. doi: 10.1007/s00134-013-3133-3. Epub 2013 Oct 25. PMID 24158410
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Mojoli F, Bouhemad B, Mongodi S, Lichtenstein D. Lung Ultrasound for Critically Ill Patients. Am J Respir Crit Care Med. 2019 Mar 15;199(6):701-714. doi: 10.1164/rccm.201802-0236CI. PMID 30372119
- [Background] Zong HF, Guo G, Liu J, Bao LL, Yang CZ. Using lung ultrasound to quantitatively evaluate pulmonary water content. Pediatr Pulmonol. 2020 Mar;55(3):729-739. doi: 10.1002/ppul.24635. Epub 2020 Jan 9. PMID 31917899
- [Background] Rouby JJ, Arbelot C, Gao Y, Zhang M, Lv J, An Y, Chunyao W, Bin D, Valente Barbas CS, Dexheimer Neto FL, Prior Caltabeloti F, Lima E, Cebey A, Perbet S, Constantin JM; APECHO Study Group. Training for Lung Ultrasound Score Measurement in Critically Ill Patients. Am J Respir Crit Care Med. 2018 Aug 1;198(3):398-401. doi: 10.1164/rccm.201802-0227LE. No abstract available. PMID 29557671
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Lichter Y, Topilsky Y, Taieb P, Banai A, Hochstadt A, Merdler I, Gal Oz A, Vine J, Goren O, Cohen B, Sapir O, Granot Y, Mann T, Friedman S, Angel Y, Adi N, Laufer-Perl M, Ingbir M, Arbel Y, Matot I, Szekely Y. Lung ultrasound predicts clinical course and outcomes in COVID-19 patients. Intensive Care Med. 2020 Oct;46(10):1873-1883. doi: 10.1007/s00134-020-06212-1. Epub 2020 Aug 28. PMID 32860069
- [Background] Dransart-Raye O, Roldi E, Zieleskiewicz L, Guinot PG, Mojoli F, Mongodi S, Bouhemad B. Lung ultrasound for early diagnosis of postoperative need for ventilatory support: a prospective observational study. Anaesthesia. 2020 Feb;75(2):202-209. doi: 10.1111/anae.14859. Epub 2019 Sep 23. PMID 31549404
- [Background] Gargani L, Lionetti V, Di Cristofano C, Bevilacqua G, Recchia FA, Picano E. Early detection of acute lung injury uncoupled to hypoxemia in pigs using ultrasound lung comets. Crit Care Med. 2007 Dec;35(12):2769-74. doi: 10.1097/01.CCM.0000287525.03140.3F. PMID 17828031
- [Background] Yin W, Zou T, Qin Y, Yang J, Li Y, Zeng X, Kang Y; Chinese Critical Ultrasound Study Group (CCUSG). Poor lung ultrasound score in shock patients admitted to the ICU is associated with worse outcome. BMC Pulm Med. 2019 Jan 3;19(1):1. doi: 10.1186/s12890-018-0755-9. PMID 30606165
- [Background] Brahier T, Meuwly JY, Pantet O, Brochu Vez MJ, Gerhard Donnet H, Hartley MA, Hugli O, Boillat-Blanco N. Lung Ultrasonography for Risk Stratification in Patients with Coronavirus Disease 2019 (COVID-19): A Prospective Observational Cohort Study. Clin Infect Dis. 2021 Dec 6;73(11):e4189-e4196. doi: 10.1093/cid/ciaa1408. PMID 32940646
- [Background] Bueno-Campana M, Sainz T, Alba M, Del Rosal T, Mendez-Echevarria A, Echevarria R, Tagarro A, Ruperez-Lucas M, Herrreros ML, Latorre L, Calvo C. Lung ultrasound for prediction of respiratory support in infants with acute bronchiolitis: A cohort study. Pediatr Pulmonol. 2019 Jun;54(6):873-880. doi: 10.1002/ppul.24287. Epub 2019 Mar 5. PMID 30838805
- [Background] Ingelse SA, Pisani L, Westdorp MHA, Almakdase M, Schultz MJ, van Woensel JBM, Bem RA. Lung ultrasound scoring in invasive mechanically ventilated children with severe bronchiolitis. Pediatr Pulmonol. 2020 Oct;55(10):2799-2805. doi: 10.1002/ppul.24974. Epub 2020 Jul 30. PMID 32696620
- [Background] Kaskinen AK, Martelius L, Kirjavainen T, Rautiainen P, Andersson S, Pitkanen OM. Assessment of extravascular lung water by ultrasound after congenital cardiac surgery. Pediatr Pulmonol. 2017 Mar;52(3):345-352. doi: 10.1002/ppul.23531. Epub 2016 Oct 14. PMID 27740725
- [Background] Cantinotti M, Giordano R, Scalese M, Marchese P, Franchi E, Viacava C, Molinaro S, Assanta N, Koestenberger M, Kutty S, Gargani L, Ait-Ali L. Prognostic Value of a New Lung Ultrasound Score to Predict Intensive Care Unit Stay in Pediatric Cardiac Surgery. Ann Thorac Surg. 2020 Jan;109(1):178-184. doi: 10.1016/j.athoracsur.2019.06.057. Epub 2019 Aug 7. PMID 31400328
- [Background] Pollack MM, Holubkov R, Funai T, Berger JT, Clark AE, Meert K, Berg RA, Carcillo J, Wessel DL, Moler F, Dalton H, Newth CJ, Shanley T, Harrison RE, Doctor A, Jenkins TL, Tamburro R, Dean JM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Simultaneous Prediction of New Morbidity, Mortality, and Survival Without New Morbidity From Pediatric Intensive Care: A New Paradigm for Outcomes Assessment. Crit Care Med. 2015 Aug;43(8):1699-709. doi: 10.1097/CCM.0000000000001081. PMID 25985385
- [Background] Senna S, Ong C, Wong JJ, Allen JC Jr, Sultana R, Lee JH. Prediction of Acquired Morbidity Using Illness Severity Indices in Pediatric Intensive Care Patients. Pediatr Crit Care Med. 2020 Nov;21(11):e972-e980. doi: 10.1097/PCC.0000000000002417. PMID 32639477
- [Background] Payen V, Jouvet P, Lacroix J, Ducruet T, Gauvin F. Risk factors associated with increased length of mechanical ventilation in children. Pediatr Crit Care Med. 2012 Mar;13(2):152-7. doi: 10.1097/PCC.0b013e3182257a24. PMID 21760567
- [Background] Farias JA, Frutos F, Esteban A, Flores JC, Retta A, Baltodano A, Alia I, Hatzis T, Olazarri F, Petros A, Johnson M. What is the daily practice of mechanical ventilation in pediatric intensive care units? A multicenter study. Intensive Care Med. 2004 May;30(5):918-25. doi: 10.1007/s00134-004-2225-5. Epub 2004 Mar 17. PMID 15029473
- [Background] Curley MA, Wypij D, Watson RS, Grant MJ, Asaro LA, Cheifetz IM, Dodson BL, Franck LS, Gedeit RG, Angus DC, Matthay MA; RESTORE Study Investigators and the Pediatric Acute Lung Injury and Sepsis Investigators Network. Protocolized sedation vs usual care in pediatric patients mechanically ventilated for acute respiratory failure: a randomized clinical trial. JAMA. 2015 Jan 27;313(4):379-89. doi: 10.1001/jama.2014.18399. PMID 25602358
- [Background] Wolfler A, Calderoni E, Ottonello G, Conti G, Baroncini S, Santuz P, Vitale P, Salvo I; SISPE Study Group. Daily practice of mechanical ventilation in Italian pediatric intensive care units: a prospective survey. Pediatr Crit Care Med. 2011 Mar;12(2):141-6. doi: 10.1097/PCC.0b013e3181dbaeb3. PMID 20351615
- [Background] Menon K, McNally D, O'Hearn K, Acharya A, Wong HR, Lawson M, Ramsay T, McIntyre L, Gilfoyle E, Tucci M, Wensley D, Gottesman R, Morrison G, Choong K; Canadian Critical Care Trials Group. A Randomized Controlled Trial of Corticosteroids in Pediatric Septic Shock: A Pilot Feasibility Study. Pediatr Crit Care Med. 2017 Jun;18(6):505-512. doi: 10.1097/PCC.0000000000001121. PMID 28406862
- [Background] Morris JV, Ramnarayan P, Parslow RC, Fleming SJ. Outcomes for Children Receiving Noninvasive Ventilation as the First-Line Mode of Mechanical Ventilation at Intensive Care Admission: A Propensity Score-Matched Cohort Study. Crit Care Med. 2017 Jun;45(6):1045-1053. doi: 10.1097/CCM.0000000000002369. PMID 28328654
- [Background] Khemani RG, Smith LS, Zimmerman JJ, Erickson S; Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: definition, incidence, and epidemiology: proceedings from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5 Suppl 1):S23-40. doi: 10.1097/PCC.0000000000000432. PMID 26035358
- [Background] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Background] Matics TJ, Sanchez-Pinto LN. Adaptation and Validation of a Pediatric Sequential Organ Failure Assessment Score and Evaluation of the Sepsis-3 Definitions in Critically Ill Children. JAMA Pediatr. 2017 Oct 2;171(10):e172352. doi: 10.1001/jamapediatrics.2017.2352. Epub 2017 Oct 2. PMID 28783810
- [Background] Leteurtre S, Duhamel A, Salleron J, Grandbastien B, Lacroix J, Leclerc F; Groupe Francophone de Reanimation et d'Urgences Pediatriques (GFRUP). PELOD-2: an update of the PEdiatric logistic organ dysfunction score. Crit Care Med. 2013 Jul;41(7):1761-73. doi: 10.1097/CCM.0b013e31828a2bbd. PMID 23685639
- [Background] Pollack MM, Patel KM, Ruttimann UE. PRISM III: an updated Pediatric Risk of Mortality score. Crit Care Med. 1996 May;24(5):743-52. doi: 10.1097/00003246-199605000-00004. PMID 8706448
- [Background] Gaies MG, Jeffries HE, Niebler RA, Pasquali SK, Donohue JE, Yu S, Gall C, Rice TB, Thiagarajan RR. Vasoactive-inotropic score is associated with outcome after infant cardiac surgery: an analysis from the Pediatric Cardiac Critical Care Consortium and Virtual PICU System Registries. Pediatr Crit Care Med. 2014 Jul;15(6):529-37. doi: 10.1097/PCC.0000000000000153. PMID 24777300